CLINICAL TRIAL: NCT04503174
Title: Control-IQ Observational (CLIO) Post-Approval Study
Acronym: CLIO
Status: Completed | Type: Observational
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: CLIO Study
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes

GROUPS / COHORTS (7):
- Pump Naive: New to insulin pump use
  Interventions: Device: t:slim X2 pump with Control-IQ technology
- 6-13 YO: Subjects between the age of 6-13 years old.
  Interventions: Device: t:slim X2 pump with Control-IQ technology
- 14-17 YO: Subjects between the age of 14-17 years old.
  Interventions: Device: t:slim X2 pump with Control-IQ technology
- Adults (18+): Subjects are 18 years old and older.
  Interventions: Device: t:slim X2 pump with Control-IQ technology
- CGM Naive: Subjects have not used CGM in the 30 days prior to enrollment.
  Interventions: Device: t:slim X2 pump with Control-IQ technology
- HbA1c more than or equal to 8.5%: Subjects have an HbA1c of more than or equal to 8.5% in the 3 months prior to enrollment.
  Interventions: Device: t:slim X2 pump with Control-IQ technology
- HbA1c less than or equal to 8.5%: Subjects have an HbA1c of less than or equal to 8.5% in the 3 months prior to enrollment.
  Interventions: Device: t:slim X2 pump with Control-IQ technology

INTERVENTIONS:
Device: t:slim X2 pump with Control-IQ technology — Real-world use

SUMMARY:
Post-approval 522 study designed to collect primarily safety data on the US FDA-cleared product, t:slim X2 insulin pump with Control-IQ technology (Control-IQ system).

DETAILED DESCRIPTION:
Post-approval study designed to collect primarily safety data on the US FDA-cleared product, t:slim X2 insulin pump with Control-IQ technology (Control-IQ system), by assessing the rate of severe hypoglycemia (SH) and diabetic ketoacidosis (DKA) during the first 12 months of use. Secondary endpoints assessing the effectiveness of this product in real-world use by assessing the impact on patients' glycemic outcomes and user experience will also be collected. The Control-IQ system will be used as intended and in accordance with FDA-approved labeling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with self-reported type 1 diabetes who have been prescribed the Control-IQ system.
* At least 6 years of age
* Using Humalog or Novolog insulin
* For females, not pregnant or planning pregnancy in the next 12 months.
* Agreement to use the t:slim X2 with Control-IQ technology, and to continue use for at least 12 consecutive months after study enrollment.
* Agree to provide HbA1c result, obtained within the 6-month period prior to enrollment.
* Ability to respond to alerts and alarms, and to provide basic diabetes self-management.
* Patients who reside full-time in the United States.
* Willingness to download the t:connect Mobile application to their Smartphone and keep it active throughout the study. Patients unable to use t:connect Mobile application must be willing to manually upload their insulin pump data to t:connect every three months and at the completion of the study.
* Subject has read, understood and agreed to participate in the study, and has electronically signed the Informed Consent Form (ICF).

Exclusion Criteria:

* Self-reported type 2 diabetes
* < 6 years of age
* Use of any glucose-lowering therapy other than Humalog or Novolog insulin
* Inability to respond to alerts and alarms, or to provide basic diabetes self-management.
* Pregnancy
* Subjects who have not signed the ICF.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects who start therapy with the Control-IQ System once the study is approved to start, that meet the indications for use and the study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3157 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Principal Investigator — Tandem Diabetes Care, Inc.
Locations (1):
- Tandem Diabetes, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Graham R, Mueller L, Manning M, Habif S, Messer LH, Pinsker JE, Aronoff-Spencer E. Real-World Use of Control-IQ Technology Is Associated with a Lower Rate of Severe Hypoglycemia and Diabetic Ketoacidosis Than Historical Data: Results of the Control-IQ Observational (CLIO) Prospective Study. Diabetes Technol Ther. 2024 Jan;26(1):24-32. doi: 10.1089/dia.2023.0341. Epub 2023 Oct 26. PMID 37782904

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3157 participants completed the baseline survey and were enrolled, but only 3061 had started closed-loop and had adequate data available for analysis.
Groups:
- All Enrolled Participants: All participants with analyzable data (minimum of 75% CGM data available for at least 21 days)
  t:slim X2 pump with Control-IQ technology: Real-world use
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 3061
Completed | 2998
Not Completed | 63

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Participants: All participants who started the monthly surveys.
  t:slim X2 pump with Control-IQ technology: Real-world use
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 3157
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29.0 [16.0 to 45.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1759
  Male | 1398
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 271
  Not Hispanic or Latino | 2819
  Unknown or Not Reported | 67
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: not mutually exclusive, not all participants answered.
  Participants
    number analyzed (Participants) | 3031
    American Indian or Alaska Native | 60
    Asian | 78
    Native Hawaiian or Other Pacific Islander | 14
    Black or African American | 184
    White | 2628
    More than one race | 0
    Unknown or Not Reported | 67
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3157

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rates of Severe Hypoglycemia (SH)
Description: Overall incidence rate of events per 100 patient years
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: events per 100 patient years
Groups:
- Prior MDI User: New to insulin pump use
  t:slim X2 pump with Control-IQ technology: Real-world use
- 6-17 YO: Subjects between the age of 6-17 years old.
  t:slim X2 pump with Control-IQ technology: Real-world use
- No Prior CGM Experience: Subjects have not used CGM in the 30 days prior to enrollment.
  t:slim X2 pump with Control-IQ technology: Real-world use
- HbA1c Greater Than or Equal to 8%: Subjects have an HbA1c greater than or equal to 8% in the 6 months prior to enrollment.
  t:slim X2 pump with Control-IQ technology: Real-world use
- HbA1c Less Than 8%: Subjects have an HbA1c of less than 8% in the 6 months prior to enrollment.
  t:slim X2 pump with Control-IQ technology: Real-world use
- Prior Pump User: Existing insulin pump user
  t:slim X2 pump with Control-IQ technology: Real-world use
- Prior CGM Experience: Subjects have used CGM in the 30 days prior to enrollment.
  t:slim X2 pump with Control-IQ technology: Real-world use
Arm/Group | Prior MDI User | 6-17 YO | Adults (18+) | No Prior CGM Experience | HbA1c Greater Than or Equal to 8% | HbA1c Less Than 8% | Prior Pump User | Prior CGM Experience
Number analyzed (Participants) | 915 | 931 | 2130 | 392 | 1295 | 1766 | 2146 | 2669
events per 100 patient years | 9.65 (36.47) | 9.31 (34.31) | 9.77 (36.97) | 7.99 (30.04) | 9.58 (37.03) | 9.66 (35.55) | 9.61 (36.06) | 9.87 (36.99)

2. Primary Outcome: Incidence Rates of Diabetic Ketoacidosis (DKA)
Description: Overall incidence rate of events per 100 patient years
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: events per 100 patient years
Arm/Group | Prior MDI User | 6-17 YO | Adults (18+) | No Prior CGM Experience | HbA1c Greater Than or Equal to 8% | HbA1c Less Than 8% | Prior Pump User | Prior CGM Experience
Number analyzed (Participants) | 915 | 931 | 2130 | 392 | 1295 | 1766 | 2146 | 2669
events per 100 patient years | 2.40 (16.69) | 1.93 (13.78) | 1.46 (13.10) | 3.57 (19.91) | 2.47 (16.50) | 0.96 (10.33) | 1.26 (11.56) | 1.37 (12.02)

3. Primary Outcome: Percent of Boluses Using the Auto Population Feature Resulting in Fewer Readings Less Than 70 mg/dL Than Those Not Using the Feature
Description: Percent of boluses using the auto population feature resulting in at least one reading less than 70 mg/dL than those not using the feature, in every pre-bolus glucose range examined.
Time Frame: 12 months
Measure: Number; unit: percentage of boluses
Groups:
- All Enrolled Participants: All participants with analyzable data
  t:slim X2 pump with Control-IQ technology: Real-world use
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 3061
percentage of boluses
  70 to 180 mg/dL Correction Bolus Results within 5 hours after bolus (with CGM auto population) | 13.18
  70 to 180 mg/dL Correction Bolus Results within 5 hours after bolus (no CGM auto population) | 14.52
  181 to 250 mg/dL Correction Bolus Results within 5 hours after bolus (with CGM auto population) | 11.06
  181 to 250 mg/dL Correction Bolus Results within 5 hours after bolus (no CGM auto population) | 15.61
  > 250 mg/dL Correction Bolus Results within 5 hours after bolus (with CGM auto population) | 10.34
  > 250 mg/dL Correction Bolus Results within 5 hours after bolus (no CGM auto population) | 13.50
  All (with CGM auto population) | 12.22
  All (no CGM auto population) | 14.60

4. Secondary Outcome: Percent Time in Range 70 - 180 mg/dL
Description: CGM measured percent time in range 70 - 180 mg/dL during 12 months of Control-IQ use
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: percentage of time
Groups:
- Overall: All subjects
  t:slim X2 pump with Control-IQ technology: Real-world use
Arm/Group | Adults (18+) | 14-17 YO | 6-13 YO | Overall
Number analyzed (Participants) | 2130 | 412 | 519 | 3061
percentage of time | 70.1 [61.0 to 78.8] | 60.9 [50.1 to 71.8] | 61.2 [52.4 to 70.5] | 67.3 [57.4 to 76.9]

5. Secondary Outcome: Percent Time Greater Than 180 mg/dL
Description: CGM measured percent time greater than 180 mg/dL during 12 months of Control-IQ use
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Adults (18+) | 14-17 YO | 6-13 YO | Overall
Number analyzed (Participants) | 2130 | 412 | 519 | 3061
percentage of time | 28.6 [19.2 to 37.8] | 37.0 [26.5 to 48.7] | 37.2 [27.5 to 46.3] | 31.4 [20.9 to 41.5]

6. Secondary Outcome: Percent Time Greater Than 250 mg/dL
Description: CGM measured percent time greater than 250 mg/dL during 12 months of Control-IQ use
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Adults (18+) | 14-17 YO | 6-13 YO | Overall
Number analyzed (Participants) | 2130 | 412 | 519 | 3061
percentage of time | 6.3 [2.8 to 12.0] | 12.8 [6.1 to 21.9] | 12.7 [7.5 to 21.0] | 8.0 [3.6 to 14.8]

7. Secondary Outcome: Percent Time Less Than 70 mg/dL
Description: CGM measured percent time less than 70 mg/dL during 12 months of Control-IQ use
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Adults (18+) | 14-17 YO | 6-13 YO | Overall
Number analyzed (Participants) | 2130 | 412 | 519 | 3061
percentage of time | 1.1 [0.5 to 2.1] | 1.0 [0.5 to 1.9] | 1.1 [0.6 to 2.2] | 1.1 [0.5 to 2.1]

8. Secondary Outcome: Percent Time Less Than 54 mg/dL
Description: CGM measured percent time less than 54 mg/dL during 12 months of Control-IQ use
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Adults (18+) | 14-17 YO | 6-13 YO | Overall
Number analyzed (Participants) | 2130 | 412 | 519 | 3061
percentage of time | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4]

9. Secondary Outcome: Diabetes Impact and Satisfaction Scale (DIDS), Satisfaction Score
Description: DIDS satisfaction score after 12 months of Control-IQ use. Score range from 0-10 with higher scores indicating better outcome.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 3061
score on a scale | 9.14 [8.29 to 9.71]

10. Secondary Outcome: Diabetes Impact and Satisfaction Scale (DIDS), Impact Score
Description: DIDS impact score after 12 months of Control-IQ use. Score range from 0 -10 with lower scores indicating better outcome.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 3061
score on a scale | 2.75 [2.0 to 4.0]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | All Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 1/3061
Serious Adverse Events (participants affected / at risk) | 14/3061
Other Adverse Events (participants affected / at risk) | 0/3061
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Participants (N=3061)
Ketosis (Endocrine disorders) | 9 (9) — Ketosis without DKA, evaluated in medical facility.
Severe Hyperglycemia (Endocrine disorders) | 3 (3) — Hyperglycemia without ketones or DKA, evaluated in medical facility.
Death (Cardiac disorders) | 1 (1) — Death secondary to complications of longstanding congenital heart disease, unrelated to blood sugar.
Chest pain (Cardiac disorders) | 1 (1) — Chest pain evaluated in emergency department unrelated to blood sugar.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT04503174/Prot_SAP_001.pdf